CLINICAL TRIAL: NCT00737113
Title: Recombinant Human Growth Hormone(RH-GH) For Accelerating Immune Reconstitution In Pediatric and Adult Patients Undergoing Allogeneic Stem Cell Transplantation
Brief Title: Recombinant Human Growth Hormone (RH-GH) For Accelerating Immune Reconstitution Post Unrelated Cord Blood Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated early due to low accrual.
Sponsor: Mitchell Horwitz, MD (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Mitchell Horwitz, MD, Assoc Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00001910
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Allogeneic Stem Cell Transplantation
Keywords: allogeneic stem cell transplantation; Engrafted; subjects
MeSH Terms: interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Genotropin (Recombinant Human Growth Hormone) — Patients will begin daily subcutaneous (SC) therapy at a starting dose of ~0.02mg/kg body weight. The study drug will continue for 90 days post enrollment.
  Other Names: rh-GH; Genotropin

SUMMARY:
The primary objective of this study is to define the safety and efficacy of recombinant human growth hormone (rh-GH, Genotropin) in a patients undergoing allogeneic transplantation.

DETAILED DESCRIPTION:
The primary objective of this study is to define the safety and efficacy of recombinant human growth hormone (rh-GH, Genotropin) in a population of patients undergoing allogeneic stem cell transplant. The secondary objectives of this study are: to evaluate the incidence of mortality due to opportunistic infections in the first 6 months, to evaluate the incidence and severity of infectious complications, to assess laboratory parameters of post-transplant immune recovery in patients on GH therapy and to determine the probability and time of neutrophil and platelet recovery on GH therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12
* <90 days following Allogeneic Transplantation.
* ANC>500/ul for 3 consecutive days.
* ≥50% donor cells in all cellular fractions tested.
* No active grade II or higher acute graft versus host disease
* Receiving ≤ 1 mg/kg/day Methylprednisolone or equivalent
* Documentation of morphologic or radiographic remission within 45 days of protocol enrollment

Exclusion Criteria:

* Patients with acute organ dysfunction requiring monitoring in the Intensive Care unit or receiving invasive interventions that may include, Hemodialysis ,CVVHD, or any form of mechanical ventilation including CPAP/BiPap at the time of starting therapy.
* Pregnant or lactating patients and those without a negative pregnancy test.
* Patients must have a life expectancy of at least 3 months.
* Patients must be HIV negative.
* Patients must not be receiving investigational agents for treatment of GVHD.
* Patients with severe veno-occlusive disease as determined by standard criteria.
* Patients with Type 1 Diabetes at the time of initiation of stem cell transplantation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To define the safety of recombinant human growth hormone (rh-GH, Genotropin) in a population of patients undergoing allogeneic transplantation | After 6, 12, 18 patients have enrolled

SECONDARY OUTCOMES:
To evaluate the incidence of mortality due to opportunistic infections in the first 6 months. | After 6, 12, and 18 patients have enrolled
To evaluate the incidence and severity of infectious complications. | After 6, 12, and 18 patients have enrolled
To assess laboratory parameters of post-transplant immune recovery in patients on GH therapy. | After 6, 12, and 18 patients enroll.
To determine the probability and time of neutrophil and platelet recovery on GH therapy. | After 6, 12, and 18 patients enroll

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States